CLINICAL TRIAL: NCT05928793
Title: The Effect of Mindfulness Practices on Positive Thinking and Stress Coping Behaviors of Earthquake Survivor Nursing Students
Brief Title: Mindfulness Practices in Earthquake Survivor Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bozok University (Other)
Collaborators: Bayburt University (Other)
Responsible Party: Principal Investigator, Betül Bal, Lecturer, Bozok University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BayburtU
Record Dates: First submitted 2023-06-24; First posted 2023-07-03 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Nursing Student; Earthquake

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness (Experimental)
  Interventions: Behavioral: mindfulness practices
- Control (No Intervention)

INTERVENTIONS:
Behavioral: mindfulness practices — Mindfulness, according to Kabat-Zinn, is "to pay attention to the present moment in a purposeful way, without judgment." Being conscious involves both attention and awareness. Conscious awareness is an observer in the background of the state of consciousness, constantly observing the inner and outer environment. It is to direct our awareness and attention to our experiences in the present moment in an accepting way with our whole body and thoughts.
  Arms: Mindfulness

SUMMARY:
Disaster; They are natural, technological or human-induced events that cause physical, economic and social losses for all or certain segments of the society, and stop or interrupt normal life and human activities. Disasters are often unavoidable. They often come suddenly and cause great suffering to the survivors. As natural disasters, especially earthquakes occur frequently in Turkey; cause human and economic losses. The 7.7 and 7.6 magnitude earthquakes in Kahramanmaraş, which occurred in February 2023 and are described as the disaster of the century, affected ten provinces, namely Gaziantep, Hatay, Osmaniye, Adıyaman, Adana, Malatya, Kilis, Diyarbakır, Şanlıurfa and Elazığ, apart from the epicenter. Nursing students who were exposed to this earthquake were adversely affected physically, psychologically, socially and economically. The psychological effects of severe traumatic events such as earthquakes are not seen in all people to the same degree. However, the reactions of individuals to traumatic situations differ in terms of both their positive thinking skills and their ability to use stress coping mechanisms.

Positive thinking is the ability to see the bright side of things and makes people more creative and constructive. Approaching events positively and evaluating them with positive thoughts also affect the quality of individuals' daily lives. Positive thinking is also linked to positive emotions, optimism, hope, joy, and happiness. Positive thinking is one of the factors that affect the quality of life and relationships. Individuals with positive thinking characteristics always keep the expectation that good events will happen, and their perspectives and approaches to events are in this direction. Individuals who have such expectations are individuals who can adapt to distressing situations or difficulties more easily than those who do not.

In this way, the individual can gain a more optimistic perspective, reduce the amount of stress he experiences and strengthen the mechanism of coping with stress.

Many studies show that; Positive thinking skills are an important factor in coping with stress and anxiety, problem solving, happiness, academic performance and even health. The fact that positive thinking skills and mechanisms for coping with stress have such an important role in human life and behavior made us think that we can also benefit from mindfulness practices in strengthening these concepts. The study was shaped within this framework and it was aimed to reveal the effect of mindfulness practices on the positive thinking skills of nursing students and the level of coping mechanisms with stress.

ELIGIBILITY:
Inclusion Criteria:

* Exposure to earthquake
* Volunteer to participate in the study

Exclusion Criteria:

* Using other relaxation techniques with a similar effect in the last 3 months and at the time of the study
* Being on medication for psychiatric reasons

Ages: 18 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2023-05-06 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-08-06 (Actual)

PRIMARY OUTCOMES:
Change in Positive Thinking Level | 8 weeks
  This form will be used to measure the positive thinking level of nursing students. In the research, it will be applied three times in total, before the application of mindfulness, after the eighth session and after the end of mindfulness practices.

SECONDARY OUTCOMES:
Change in the Level of Coping with Stress for Nursing Students | 8 weeks
  This form will be used to measure the level of coping with stress in nursing students. In the research, it will be applied three times in total, before the application of mindfulness, after the eighth session and after the end of mindfulness practices.

CONTACTS AND LOCATIONS:
Locations (1):
- Betül, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided